CLINICAL TRIAL: NCT05881031
Title: Single Site Feasibility and Safety Study of Home Initiation of Noninvasive Positive Pressure Ventilation in Children With Medical Complexity
Brief Title: Home Initiation of Noninvasive Positive Pressure Ventilation in Children With Medical Complexity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000080480
Record Dates: First submitted 2023-05-01; First posted 2023-05-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Sleep-Disordered Breathing
Keywords: noninvasive ventilation; home mechanical ventilation
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: This will be a 12-week, open-label feasibility study of a pragmatic, two-arm parallel-group, randomized controlled trial with 1:1 allocation of children newly initiating NiPPV that compares home NiPPV initiation to usual care of initiating NiPPV in a one-night in-hospital polysomnogram.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Standard of care is NiPPV initiation during a one-night, in-hospital PSG, during which NiPPV settings are titrated during the night by a PSG technologist to determine optimal settings according to current international guidelines. Once NiPPV equipment is obtained and NiPPV is used at home (time 0), NiPPV setting changes may occur at 1, 4, and 12 weeks when participants are contacted by the respiratory therapist. Additional titration of NiPPV settings may be guided by reported participant symptoms and comfort, as per standard of care.
- Home Initiation of NiPPV (Experimental): NiPPV settings will be titrated during an awake NiPPV trial by the respiratory therapist. Once NiPPV equipment is obtained and NiPPV is used at home (time 0), further titration of the NiPPV settings will occur on an outpatient basis guided by remote telemonitoring and home overnight oximetries at 1, 4, and 12 weeks. Additional titration of NiPPV settings may be guided by reported participant symptoms and comfort, as per standard of care. Participants will complete an in-hospital PSG after 12 weeks, during which NiPPV settings are titrated during the night by a PSG technologist to determine optimal settings according to current international guidelines.
  Interventions: Other: Home Initiation of NiPPV

INTERVENTIONS:
Other: Home Initiation of NiPPV — Initiation of NiPPV in the home environment through the utilization of an awake NiPPV titration, oximetries, and telemonitoring.
  Arms: Home Initiation of NiPPV

SUMMARY:
Children with medical complexity (CMC) often have trouble breathing at night and need to use a breathing machine. This breathing machine is called noninvasive positive pressure ventilation (NiPPV). The use of NiPPV has been shown to improve quality of life and survival in children. Before it is used, NiPPV must first be tested to see what the correct 'machine settings' are for each child. This is usually done in the sleep laboratory at the hospital during a one-night stay. However, sleep studies in the hospital are disruptive and hard for CMC and their families because of the new environment and limited access to the equipment, supplies, comfort items and the routine their child has at home. Patients and families would prefer to start NiPPV at home but there needs to be more research on this to make sure it is possible and safe. This study will evaluate a new model of care to start NiPPV in the home. CMC aged 5-17 years old and starting NiPPV will be assigned at random, like a coin toss, to start NiPPV in the home or to start NiPPV in the sleep laboratory. The investigators will assess the feasibility and safety of the two ways to start NiPPV. This study will be the first step towards developing a study to evaluate if home NiPPV starts are effective. Starting NiPPV at home has the potential to improve the use of NiPPV (ie early adherence predicts long-term use) resulting in both medical benefits as well as improved quality of life for CMC and their families.

DETAILED DESCRIPTION:
Children with medical complexity (CMC) are increasingly prescribed noninvasive positive pressure ventilation (NiPPV) for chronic respiratory failure. In our clinical experience, patients and families would prefer NiPPV initiation in the home environment but this is not standard of care. This proposal will evaluate the feasibility and safety of an innovative model of care for NiPPV initiation in the home environment utilizing remote telemonitoring compared to usual care which is in-hospital polysomnography (PSG) laboratory-based initiation.

The incidence of CMC requiring NiPPV is exponentially growing. NiPPV effectively corrects abnormal gas exchange, improves sleep quality, and reduces symptoms of chronic respiratory failure. The use of NiPPV has been associated with increased survival and improved health-related quality of life (HRQOL). To ensure effectiveness, NiPPV must be used for all periods of sleep and settings must be individually-titrated. Unfortunately, poor adherence results in many CMC being undertreated for chronic respiratory failure. Successful NiPPV initiation is critical because early negative experiences are commonly reported barriers to adherence6 and early usage predicts longer term use. Standard of care is the initiation and titration of NiPPV during a one-night in-hospital PSG. A PSG is challenging for CMC and families due to their medical fragility and lasting effects of travel and a disrupted routine, the significant amount of equipment and supplies that must be brought to the study as well as the financial implications and additional psychosocial stress for caregivers. In addition, negative experiences with NiPPV may be exacerbated by introduction of the therapy in an unfamiliar PSG laboratory with burdensome monitoring. Furthermore, a one-night PSG provides limited sleep data that may not be representative of dynamic and variable sleeping patterns that occur in the comfort of one's home.

Recent technological advances in remote NiPPV monitoring coupled with a shift to virtual care models has enabled a patient and family centered opportunity to bypass the PSG laboratory and initiate NiPPV at home. Remote NiPPV monitoring extends data collection beyond discrete health care encounters and provides real-time data on adherence and efficacy that can be wirelessly transmitted to facilitate setting adjustment by clinicians. Home NiPPV initiation is increasingly being requested by patients and caregivers. The potential benefits of this innovative care model include increasing patient and family empowerment, improving the delivery of high quality patient-centred care at home, and optimizing NiPPV use. Although there is growing data in the adult population to support home NiPPV initiation via telemonitoring, this cannot be simply extrapolated to CMC. There are key differences in the etiology and manifestation of chronic respiratory failure in CMC compared to adults. Furthermore, family caregivers play an important role in NiPPV acceptance and adherence.

Canadian guidelines acknowledge the lack of evidence for the setting in which NiPPV is initiated. Home NiPPV initiation in CMC is a novel model of care that may result in large health system impacts, but requires a feasibility study before embarking on a large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-17 years old
2. Newly prescribed NiPPV
3. Tolerated awake NiPPV trial
4. Provides informed consent

Exclusion Criteria:

1. Cardiac disease at risk of hemodynamic instability with NiPPV initiation (eg cardiac dysfunction (ejection fraction <45%), pulmonary hypertension (mean pulmonary artery pressure ≥ 20 mmHg on right heart catheterization or suggestive echocardiogram findings in the opinion of a pediatric cardiologist), or single ventricle)
2. At high risk of complications with NiPPV in the opinion of the child's physician (eg pneumothorax and aspiration risk)
3. Severe sleep disordered breathing with peak CO2 ≥ 60mmHg or apnea-hypopnea index (AHI)≥ 30/hr (AHI measures the number of respiratory events per hour)
4. Participation in concurrent research study that may affect NiPPV adherence (proposed primary outcome of full study)
5. Exclusion of study participants if the caregiver or participant is not English speaking

Ages: 60 Months to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rate | 2 years
  Feasibility outcome.
  The recruitment rate is the proportion of eligible people recruited to the trial. This is the number of people randomised divided by the number of people eligible.
  The retention rate is the proportion of randomised people who complete follow up at 3 months (end of trial).
Proportion of eligible patients randomized | 2 years
  Feasibility outcome. Proportion of eligible participants who are recruited to the study and randomized
Proportion of patients that crossover based on safety criteria | 2 years
  Safety outcome. Proportion of patients in the intervention arm who crossover to the control arm based on pre-specified monitoring criteria

SECONDARY OUTCOMES:
Mean minutes of nightly NiPPV usage | 12 weeks
  Proposed trial outcome. Adherence will be determined adjectively using ventilator download data.
Proxy-reported Psychological Scale (percentage rank) | 12 weeks
  Proposed trial outcome. The proxy-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating a "dissatisfaction with life".
Proxy-reported Psychological Scale (percentage rank) | 4 weeks
  Proposed trial outcome. The proxy-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating a "dissatisfaction with life".
Proxy-reported Psychological Scale (T-value) | 12 weeks
  Proposed trial outcome. The proxy-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The T-values have a mean of 50 and standard deviation of 10. Higher T-values indicate a higher quality of life.
Proxy-reported Psychological Scale (T-value) | 4 weeks
  Proposed trial outcome. The proxy-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The T-values have a mean of 50 and standard deviation of 10. Higher T-values indicate a higher quality of life.
Self-Reported Psychological Scale (percentage rank) | 12 weeks
  Proposed trial outcome. The self-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating a "dissatisfaction with life".
Self-Reported Psychological Scale (percentage rank) | 4 weeks
  Proposed trial outcome. The self-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The percentage rank range is 0-100, with lower scores indicating a "dissatisfaction with life".
Self-Reported Psychological Scale (T-value) | 12 weeks
  Proposed trial outcome. The self-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The T-values have a mean of 50 and standard deviation of 10. Higher T-values indicate a higher quality of life.
Self-Reported Psychological Scale (T-value) | 4weeks
  Proposed trial outcome. The self-reported Psychological Scale from the KIDSCREEN-52 questionnaire will be used. The T-values have a mean of 50 and standard deviation of 10. Higher T-values indicate a higher quality of life.
Caregiver reported Sense of Mastery | 12 weeks
  Proposed trial outcome. The Pearlin Mastery Scale will be used to measure parental mastery. Scores range from 7 to 28, with higher scores indicating greater levels of mastery.
Caregiver reported Sense of Mastery | 4 weeks
  Proposed trial outcome. The Pearlin Mastery Scale will be used to measure parental mastery. Scores range from 7 to 28, with higher scores indicating greater levels of mastery.
Patient and family study experience, preference of intervention and barriers | 12 weeks
  Feasibility and acceptability outcome. Based on optional qualitative interview with participant and/or caregiver after completion of study procedures.
Difference in expiratory positive airway pressure based on home NiPPV titration and PSG titration in the intervention arm | 12 weeks
  Safety outcome. Comparison of final NiPPV settings at 12 weeks in the intervention arm and PSG prescribed NiPPV settings at 12 weeks and beyond.
Difference in inspiratory positive airway pressure based on home NiPPV titration and PSG titration in the intervention arm | 12 weeks
  Safety outcome. Comparison of final NiPPV settings at 12 weeks in the intervention arm and PSG prescribed NiPPV settings at 12 weeks and beyond.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Amin, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada